CLINICAL TRIAL: NCT01166724
Title: Renal Allograft Function and Histology Following Switching From A Tacrolimus to Sirolimus (SRL)-Based Immunosuppression- Clinical and Mechanistic Impact
Brief Title: Renal Allograft Function and Histology Following Switching From A Tacrolimus to Sirolimus (SRL)-Based Immunosuppression-
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Collaborator stopped study
Sponsor: The Cleveland Clinic (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09-702
Record Dates: First submitted 2010-07-20; First posted 2010-07-21 (Estimated); Results first posted 2017-06-07 (Actual); Last update posted 2017-06-07 (Actual); Status verified 2017-02

CONDITIONS: Kidney Transplant
Keywords: Kidney transplant
MeSH Terms: interventions — Sirolimus; Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sirolimus (Active Comparator): patients will be switched from Tacrolimus to Sirolimus
  Interventions: Drug: Sirolimus; Drug: Tacrolimus
- Tacrolimus (No Intervention): Patient will stay on Tacrolimus

INTERVENTIONS:
Drug: Sirolimus — Tacrolimus to Sirolimus
  Arms: Sirolimus
Drug: Tacrolimus — dosage per trough level
  Arms: Sirolimus

SUMMARY:
The investigators hypothesize that Tacrolimus (Tac) withdrawal from a Tac, MMF and steroid based triple therapy regimen leads to long term improved/stabilized graft function (glomerular filtration rate, GFR) primarily as a consequence of halting CNI-induced fibrogenetic processes that mediate loss of functioning renal tissue. The investigators further hypothesize that the underlying fibrotic mechanism is mediated by pathophysiologic processes that promote epithelial to mesenchymal transition (EMT) (mediated by TGF- ƒÒ) and that early therapeutic intervention may reverse this process (mediated by BMP-7)4.

To address these hypotheses the investigators propose the following clinical and mechanistic aims:

The investigators will test the hypothesis that switching from Tac to SRL in a Tac based triple therapy regimen with MMF and steroids in living and or deceased donor renal transplant recipients leads to improvement in allograft structure and function at 2 years post-transplantation.

The investigators will test this hypothesis in an open label controlled trial where stable renal allograft recipients on Tac, MMF, prednisone maintenance immunosuppression will undergo renal biopsy at 3-4 months post-transplantation and will be randomized to either a) Remain on Tac, MMF and prednisone (CNI-maintenance) or b) switch the Tac to SRL and continue MMF and prednisone. The investigators will then compare biopsy derived measures of allograft fibrosis (CADI, Sirius Red, Banff Chronicity Index) and GFR in the two groups

DETAILED DESCRIPTION:
We will test this hypothesis in an open label controlled trial where stable renal allograft recipients on Tac, MMF, prednisone maintenance immunosuppression will undergo renal biopsy at 3-4 months post-transplantation and will be randomized to either a) Remain on Tac, MMF and prednisone (CNI-maintenance) or b) switch the Tac to SRL and continue MMF and prednisone. We will then compare biopsy derived measures of allograft fibrosis (CADI, Sirius Red, Banff Chronicity Index) and GFR in the two groups

ELIGIBILITY:
Inclusion Criteria:

1. Absence of clinical acute rejection in post-transplant period preceding randomization
2. HLA-mismatched solitary first and second kidney transplant recipients
3. Absence of any degree of rejection (Banff 2007) on renal biopsy at 3-6 months(+/- 2 months) post-transplant.
4. Absence of post-transplant donor-specific antibody

Exclusion Criteria:

1. HLA-identical transplants
2. Contraindication or inability to undergo renal biopsy, like previous complications due to biopsies, anticoagulation, active infection, etc.
3. Positive flow cross match, sensitized recipient, presence of donor-specific antibody.
4. Rejection episode after transplantation, either cellular or humoral on for cause or renal biopsy.
5. Rejection present on pre-randomization renal biopsy.
6. Proteinuria greater than 0.3 gram/day
7. Native kidney disease biopsy proven or likely glomerulonephritis, primary or recurrent FSGS, MPGN or primary or recurrent membranous GN.
8. Hypertriglyceridemia > 400 mg/dL (treated), LDL cholesterol > 160 mg/dL while on optimal treatment.
9. WBC < 2000/mm3, ANC < 1000 mm3, Platelet count < 100,000 mm3
10. Active wound issues.
11. Primary non-function.
12. Active BKV or CMV disease.
13. Evidence of recurrent disease.
14. Active infection
15. Pregnancy
16. Women of childbearing potential unable or unwilling to use birth control during the study.
17. e GFR ≤ 40 ml/ min at screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2010-07; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: T Srinivas, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Sirolimus: patients will be switched from Tacrolimus to Sirolimus
  Sirolumus: Tacrolimus to Sirolimus
  Tacrolimus: dosage per trough level
Period: Overall Study
Arm/Group | Sirolimus | Tacrolimus
Started | 7 | 5
Completed | 0 | 0
Not Completed | 7 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sirolimus | Tacrolimus | Total
Number analyzed (Participants) | 7 | 5 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 5 | 11
  >=65 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 5 | 2 | 7
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Biopsy-derived Measures of Fibrosis
Description: The primary analyses will compare biopsy-derived measures of fibrosis in the Tac-maintenance and SRL groups using the t-test.
Time Frame: 12 months
Population: Early termination; Sponsor discontinued the study for corporate reasons. No data analyzed. Data were not collected and the outcome measure was not analyzed.
Arm/Group | Sirolimus | Tacrolimus
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Change in iGFR
Description: We will also compare the change in iGFR (as well as estimated GFR) from time of conversion to 12 and 24 months of follow up by paired t-test between groups.
Time Frame: 12 months
Population: as for outcome 1
Arm/Group | Sirolimus | Tacrolimus
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Sirolimus | Tacrolimus
Serious Adverse Events (participants affected / at risk) | 2/7 | 0/5
Other Adverse Events (participants affected / at risk) | 4/7 | 0/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sirolimus (N=7) | Tacrolimus (N=5)
Pruritus; Pancreatitis (Endocrine disorders) | 1 | 0
ER Admit: Fever, Vomitting (General disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sirolimus (N=7) | Tacrolimus (N=5)
ER Admit: Fever, Vomitting (General disorders) | 1 | 0
Food Poisoning (Gastrointestinal disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Fever, Cough (General disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
Early termination; Sponsor discontinued the study for corporate reasons. No data analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes